CLINICAL TRIAL: NCT02324452
Title: Safety, Feasibility and Cost-effectiveness of Genotype-directed Individualized Dosing of Fluoropyrimidines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14DPD; 2014-005064-15 (EudraCT Number)
Record Dates: First submitted 2014-12-09; First posted 2014-12-24 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- heterozygous carrier of DPYD variant (Experimental): Patients screened for four single nucleotide polymorphisms (SNPs) in DPYD (DPYD*2A, c.2846A>T, c.1236G>A/HapB3 and DPYD*13) that are found to be heterozygous for one of these SNPs
  Interventions: Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil)
- wild type for DPYD (Experimental): Patients screened for four single nucleotide polymorphisms (SNPs) in DPYD (DPYD*2A, c.2846A>T, c.1236G>A/HapB3 and DPYD*13) that are found to be wild type for these SNPs
  Interventions: Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil)

INTERVENTIONS:
Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil) — Patient that are a heterozygous carrier of a DPYD variant will receive a reduced dosage of capecitabine or 5-fluorouracil (25-50% reduction, depending on which SNP is identified). The dose will be titrated in subsequent cycles, to achieve maximal safe exposure. Patients that are wild type (not carrying any of the for DPYD variants) will receive a normal (full) dose.
  Other Names: Xeloda; Capecitabine; 5-fluorouracil; fluorouracil; 5-FU

SUMMARY:
In this study it will be determined whether the rate of severe toxicity associated with fluoropyrimidine treatment (capecitabine or 5-fluorouracil) can be significantly diminished by individualized dosing of fluoropyrimidines based on upfront genotypic assessment of dihydropyrimidine dehydrogenase (DPD) deficiency.

In addition to the genotyping, the DPD phenotype of all patients will be determined by measuring the baseline dihydrouracil/uracil (DHU/U) ratio, in order to investigate whether phenotype-guided treatment can further improve patient safety. In a subgroup of patients, other phenotyping methods will be tested: measuring the plasma levels of uracil after a uracil test dose and a uracil breath test after a dose of [2-13C] -labeled uracil. To validate these tests, these phenotyping results will be compared with the results of a DPD activity assay (which measures DPD enzyme activity in peripheral blood mononuclear cells), which is considered the gold standard in measuring DPD phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed malignancy for which treatment with a fluoropyrimidine is considered to be in the patient's best interest
2. Age ≥ 18 years
3. Able and willing to give written informed consent
4. WHO performance status of 0, 1 or 2
5. Life expectancy of at least 12 weeks
6. Able to swallow and retain oral medication
7. Able and willing to undergo blood sampling for pharmacogenetic and phenotyping analysis
8. Minimal acceptable safety laboratory values (ANC, platelet count, hepatic function, renal function)

Additional inclusion criteria for patients in subgroup of study:

1. Able and willing to undergo blood sampling and breath sampling at several time points
2. Able and willing to receive uracil for the test dose assay
3. Able and willing to receive [2-13C] -labeled uracil for the breath test

Exclusion Criteria:

1. Prior treatment with fluoropyrimidines
2. Patients with known substance abuse, psychotic disorders, and/or other diseases expected to interfere with study or the patient's safety
3. Women who are pregnant or breast feeding
4. Both men and women who refuse to use reliable contraceptive methods throughout the study (adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms)
5. Patients with a homozygous polymorphic genotype or compound heterozygous genotype for DPYD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1103 (Actual)
Dates: Start 2015-03; Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of severe treatment-related toxicity (CTC grade 3 to 5) | patients will be followed during fluoropyrimidine treatment, expected average of 1 year
  The incidence of severe treatment-related toxicity (CTC grade 3 to 5) in patients carrying DPYD variants compared to wild type patients and compared to a historical cohort of DPYD heterozygous patients treated with a full dose of fluoropyrimidines

SECONDARY OUTCOMES:
Cost-effectiveness: medical costs that are made during fluoropyrimidine treatment seen from a health care perspective | patients will be followed during fluoropyrimidine treatment, expected average of 1 year
  Costs in the group where dose individualization of fluoropyrimidines based on upfront genotyping is performed is compared to a historic cohort without dose individualization. Costs include costs for genotyping, fluoropyrimidine drug therapy and costs related to adverse events.
DPD phenotype, defined as deficient or not deficient | Prior to start of fluoropyrimidine treatment of the patient (pre dose)
  Several phenotyping tests that assess DPD enzyme activity will be compared and clinical sensitivity, specificity, positive predictive value and negative predictive value of each test will be determined
Assessment of pharmacokinetics: Such profile parameters will include Cmax, Tmax, AUC and elimination half-life | At first week of start of fluoropyrimidine treatment of the patient
  In patients with heterozygous DPYD mutations the plasma levels of capecitabine, 5-FU and metabolites will be determined to assess the pharmacokinetic (PK) profile in these patients given reduced doses of capecitabine and 5-FU

CONTACTS AND LOCATIONS:
Overall Officials: JHM Schellens, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (17):
- Netherlands (17):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Wilhelmina Hospital Assen, Assen
  - Amphia Hospital, Breda
  - Reinier de Graaf Hospital, Delft
  - Deventer Hospital, Deventer
  - Hospital Gelderse Vallei, Ede
  - Catharina Hospital, Eindhoven
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Laurentius Hospital, Roermond
  - Bravis Hospital, Roosendaal
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Haga Hospital, The Hague
  - Medical Center Haaglanden, The Hague
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Knikman JE, Lopez-Yurda M, Meulendijks D, Deenen MJ, Schellens JHM, Beijnen J, Cats A, Guchelaar HJ. A Nomogram to Predict Severe Toxicity in DPYD Wild-Type Patients Treated With Capecitabine-Based Anticancer Regimens. Clin Pharmacol Ther. 2024 Feb;115(2):269-277. doi: 10.1002/cpt.3100. Epub 2023 Nov 29. PMID 37957132
- [Derived] Knikman JE, Wilting TA, Lopez-Yurda M, Henricks LM, Lunenburg CATC, de Man FM, Meulendijks D, Nieboer P, Droogendijk HJ, Creemers GJ, Mandigers CMPW, Imholz ALT, Mathijssen RHJ, Portielje JEA, Valkenburg-van Iersel L, Vulink A, van der Poel MHW, Baars A, Swen JJ, Gelderblom H, Schellens JHM, Beijnen JH, Guchelaar HJ, Cats A. Survival of Patients With Cancer With DPYD Variant Alleles and Dose-Individualized Fluoropyrimidine Therapy-A Matched-Pair Analysis. J Clin Oncol. 2023 Dec 10;41(35):5411-5421. doi: 10.1200/JCO.22.02780. Epub 2023 Aug 28. PMID 37639651
- [Derived] Henricks LM, Lunenburg CATC, de Man FM, Meulendijks D, Frederix GWJ, Kienhuis E, Creemers GJ, Baars A, Dezentje VO, Imholz ALT, Jeurissen FJF, Portielje JEA, Jansen RLH, Hamberg P, Ten Tije AJ, Droogendijk HJ, Koopman M, Nieboer P, van de Poel MHW, Mandigers CMPW, Rosing H, Beijnen JH, Werkhoven EV, van Kuilenburg ABP, van Schaik RHN, Mathijssen RHJ, Swen JJ, Gelderblom H, Cats A, Guchelaar HJ, Schellens JHM. DPYD genotype-guided dose individualisation of fluoropyrimidine therapy in patients with cancer: a prospective safety analysis. Lancet Oncol. 2018 Nov;19(11):1459-1467. doi: 10.1016/S1470-2045(18)30686-7. Epub 2018 Oct 19. PMID 30348537
- [Derived] Jacobs BA, Deenen MJ, Pluim D, van Hasselt JG, Krahenbuhl MD, van Geel RM, de Vries N, Rosing H, Meulendijks D, Burylo AM, Cats A, Beijnen JH, Huitema AD, Schellens JH. Pronounced between-subject and circadian variability in thymidylate synthase and dihydropyrimidine dehydrogenase enzyme activity in human volunteers. Br J Clin Pharmacol. 2016 Sep;82(3):706-16. doi: 10.1111/bcp.13007. Epub 2016 Jun 3. PMID 27161955